CLINICAL TRIAL: NCT04168866
Title: Operative Versus Non-Operative Management for Appendicitis With Abscess or Phlegmon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000026799; No NIH funding (Other: 10.11.23)
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Drainage; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery (Experimental): Patients who choose operations will have surgery performed to remove the appendix laparoscopically, through 3 or 4 small incisions. All patients in the operative group will receive standard perioperative antibiotics. They will also have the abscess(es) drained during the same surgery if there is one present. In some cases, the operation may be too difficult to perform laparoscopically, so an open appendectomy will be performed, involving a longer incision to remove the appendix. In some cases, both laparoscopic and open are performed. The surgeon may also choose to remove a section of the intestine with the appendix or perform additional procedures.
  Interventions: Procedure: Operative management
- Non-operative management (Active Comparator): If a patient chooses non-operative management and if an abscess is present and amenable to percutaneous drainage this will be performed. If there is no abscess or it is not amenable to drainage antibiotics alone will be provided.
  Interventions: Other: Drainage or antibiotics

INTERVENTIONS:
Procedure: Operative management — Surgery for computer tomography (CT)-proven complicated appendicitis with phlegmon or abscess.
  Arms: Surgery
Other: Drainage or antibiotics — If an abscess is present and amenable to percutaneous drainage this will be performed. If there is no abscess or it is not amenable to drainage antibiotics alone will be provided.
  Arms: Non-operative management

SUMMARY:
The investigators aim to determine if early operative intervention is superior to non-operative management for adult patients with computerized tomography (CT)-proven complicated appendicitis with phlegmon or abscess.

DETAILED DESCRIPTION:
Complicated appendicitis with abscess or phlegmon represents a challenging problem to emergency general surgeons, and the preferred treatment remains controversial. A variety of therapies have been recommended including early operative intervention, delayed operative intervention, and non-operative management. Recently, a prospective randomized controlled trial from a single center was conducted in Finland comparing operative and non-operative management of appendiceal abscess. Patients managed in the operative arm were found to have a shorter length of stay, fewer re-admissions, and fewer additional interventions than those managed in the non-operative group, but there is no high-quality randomized control trial conducted in the United States to support this. The investigators, therefore plan to carry out a multi-center, patient choice study comparing operative and non-operative management of complicated appendicitis with abscess or phlegmon in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Complicated appendicitis with presumed perforation on (computer tomography) CT scan AND phlegmon or abscess greater than 2 centimeter (cm).

Exclusion Criteria:

1. Antibiotic therapy greater than 24 hours prior to considering for enrollment.
2. Attempted drainage before randomization
3. Pregnancy
4. Antibiotic allergy requiring the use of something other than a beta-lactam or quinolone based therapy.
5. Previous major intra-abdominal surgery by laparotomy
6. Hospitalization within 2 weeks of randomization
7. Presence of septic shock on admission.
8. Mechanical ventilation
9. Acute renal failure requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of hospital days | Within 60 days of randomization.
  This includes all hospital days during the initial stay and any readmission.

SECONDARY OUTCOMES:
Need for additional intervention for appendicitis | Within one year of the index admission.
  Percutaneous drainage, unplanned operative intervention.
Intra-abdominal abscess | More than 7 days after index admission but within 60 days of randomization.
Failed attempted procedure. | Within 60 days of randomization.
  Conversion from laparoscopic to open surgery, conversion from non-operative to operative management, percutaneous drainage not possible or unsuccessful.
Complications | Within 60 days of randomization.
  Defined by National Surgical Quality Improvement Program criteria.
Number of interventions for abscess | Within 60 days of randomization.
Need for bowel resection. | Within 60 days of randomization.
Need for bowel resection | Within 60 days of randomization.
Occurrence of delayed appendectomy | Within one year of index admission.
Recurrence | Within one year of index admission.
Presence of malignancy in any resected specimen | Within one year of index admission.
Days of disability | Within 60 days of randomization.
  Days away from work or school.
Gastrointestinal (GI) quality of life | 30 days after randomization.
  This outcome will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Gastrointestinal Symptoms Scale. This scale includes 8 subscales of which the investigators will use 6 for a maximum of 41 items, though usually less due to skip logic. Each item is measured on a 5-point scale. Items are summed by subscale and converted to a final score by a computer algorithm. A higher score indicates greater symptom severity and lower quality of life.
GI quality of life | 60 days after randomization.
  This outcome will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Gastrointestinal Symptoms Scale. This scale includes 8 subscales of which the investigators will use 6 for a maximum of 41 items, though usually less due to skip logic. Each item is measured on a 5-point scale. Items are summed by subscale and converted to a final score by a computer algorithm. A higher score indicates greater symptom severity and lower quality of life.
GI quality of life | One year after randomization.
  This outcome will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Gastrointestinal Symptoms Scale. This scale includes 8 subscales of which the investigators will use 6 for a maximum of 41 items, though usually less due to skip logic. Each item is measured on a 5-point scale. Items are summed by subscale and converted to a final score by a computer algorithm. A higher score indicates greater symptom severity and lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mentula P, Sammalkorpi H, Leppaniemi A. Laparoscopic Surgery or Conservative Treatment for Appendiceal Abscess in Adults? A Randomized Controlled Trial. Ann Surg. 2015 Aug;262(2):237-42. doi: 10.1097/SLA.0000000000001200. PMID 25775072